CLINICAL TRIAL: NCT02826031
Title: A Multi-center, Randomized, Open-label, Parallel-arm Controlled Study Comparing Demand-based Monotherapy of Non-steroidal Anti-inflammatory Drug (NSAID) vs. Demand-based NSAID Combined With Sodium Hyaluronate Injection in the Treatment of Chinese Patients With Mild to Moderate Knee Osteoarthritis
Brief Title: Clinical Study of Artz in the Treatment of Knee Osteoarthritis
Acronym: Artz
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kunming Baker Norton Pharmaceutical Sales Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTZ2013PMS01
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
Keywords: Sodium Hyaluronate; mild to moderate knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

ARMS (2):
- Sodium Hyaluronate Injection + DICL-SR (Experimental): Each syringe (2.5mL) contains 25mg of sodium hyaluronate, and one Artz® will be administered via intra-articular injection into the target knee at the baseline and Weeks 1, 2, 3 and 4 respectively for the combination group.
  From the run-in period to the end of study, both groups will receive DICL-SR 75mg, which is administered on demand for treatment of knee pain. If the knee pain is relieved or has disappeared, DICL-SR may be withdrawn. However, if the pain occurs again and requires treatment, the drug may be resumed. If a dose of 75mg daily fails to control the knee pain, it may be increased to the maximum dose 150mg daily upon the approval of the investigator, that is, 75mg bis in die（BID） daily
  Interventions: Drug: Sodium Hyaluronate Injection; Drug: DICL-SR
- DICL-SR (Active Comparator): From the run-in period to the end of study, both groups will receive Diclofenac Sodium Sustained-release Tablets(DICL-SR) 75mg, which is administered on demand for treatment of knee pain. If the knee pain is relieved or has disappeared, DICL-SR may be withdrawn. However, if the pain occurs again and requires treatment, the drug may be resumed. If a dose of 75mg daily fails to control the knee pain, it may be increased to the maximum dose 150mg daily upon the approval of the investigator, that is, 75mg bis in die（BID daily）. A subject is allowed to withdraw from this study prematurely if unable to tolerate the adverse effects.
  Interventions: Drug: DICL-SR

INTERVENTIONS:
Drug: Sodium Hyaluronate Injection
  Arms: Sodium Hyaluronate Injection + DICL-SR
Drug: DICL-SR

SUMMARY:
This is a multi-center, randomized, open-label, parallel-arm phase IV clinical study, for which a total of 300 patients with mild to moderate knee osteoarthritis will be enrolled. In the first 4 weeks (run-in period), the subjects will receive on-demand treatment with Diclofenac Sodium Sustained Release Tablets (DICL-SR) 75mg, quaque die（QD）. After the run-in period, the subjects, if their knee pain has not worsened to a level requiring surgical treatment, will be randomized to two groups in 1:1 ratio: one group receiving Artz® via intra-articular injection (once weekly, for 5 consecutive weeks) in combination with DICL-SR 75mg,quaque die（QD）, for 12 consecutive weeks on demand. The other group receiving DICL-SR 75mg alone,quaque die（QD）, for 12 consecutive weeks on demand. DICL-SR 75mg quaque die（QD） may be administered to the subjects of both groups on demand as long as they have a knee pain. If the knee pain has disappeared, this drug may be withdrawn. However, if the pain occurs again and requires treatment, oral administration of DICL-SR may be resumed. A subject is allowed to withdraw from this study prematurely if unable to tolerate the adverse effects.

A total of 8 visits have been scheduled for this study, including Visit 1/screening period (Week -4), Visit 2/baseline (Week 0), Visit 3 (Week 1), Visit 4 (Week 2), Visit 5 (Week 3), Visit 6 (Week 4), Visit 7 (Week 8) and Visit 8 (Week 12).

A total of 300 subjects will participate in this study at 6 to 8 centers in China, and patient enrollment is expected to take up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Chinese subjects, at age≥18, either gender, diagnosed with osteoarthritis of the target knee and Kellgren-Lawrence (KL) classification Grade 1~3, as evidenced by X-ray examination in the last 3 months (mild to moderate narrowing of joint space and / or marked osteophytes of tibiofemoral joint space)
2. Persist pain of the target knee after exercise, weight loss and physical therapy;
3. A baseline WOMAC A1 score for the target knee rated at 40-90mm (moderate to severe walk-associated pain) on 100mm Visual analogue scale(VAS); Able to understand and sign the Informed Consent Form (ICF) that has already been approved by the Independent Ethics Committee (IEC) Note: the informed consent may also be given by the duly authorized representative of the subject.

Exclusion Criteria:

1. A diagnosis of bilateral knee osteoarthritis;
2. Clinically significant (requiring surgery) valgus or varus deformity of the knee joint, ligamentous laxity or unstable meniscus;
3. Complicated by inflammation or any other disease /condition (e.g., rheumatic arthritis, metabolic bone disease, psoriasis, gout, pseudogout, chondrocalcinosis, etc.) that may affect the knee joint;
4. A history of septicemia, clinically considered sub-acute infection of the target knee joint;
5. A history of surgery on the target knee (in the last 6 months);
6. A history of asthma, urticaria or allergy after use of aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs);
7. Severe hepatic or renal disease or hepatic /renal failure;
8. Any unscheduled surgery on the lower limb;
9. Clinically significant lower venous or lymphatic obstruction;
10. Clinically significant obvious exudation or inflammation of the target knee;
11. Skin disorders or infection at the injection site;
12. Pregnant or lactating women;
13. Known allergy to guanylin and / or any active ingredient or excipient of hyaluronic acid-based injection / diclofenac sodium;
14. Treatment with any hyaluronic acid (HA) or its derivatives for the target knee within six months before this trial;
15. Intra-articular (IA) injection of steroids into the target knee within 3 months before this trial;
16. Presence of any contraindication to IA injection, e.g., patients who are receiving anti-coagulation therapy or clinically have potential coagulation disorders (e.g., hepatic disease);
17. Presence of any clinically significant disease (e.g., significant mental or nervous disorders, alcohol/drug abuse), unstable/poorly controlled diseases, or other factors, which may affect their evaluation or participation in this study in the investigator's judgment
18. Perioperative pain associated with coronary artery bypass surgery (CABG);
19. A history of gastrointestinal bleeding or perforation following use of NSAIDs;
20. Presence of active gastrointestinal ulcer /bleeding, or a past history of recurrent ulcer/bleeding; Chief complaint complicated by pain beyond the target knee,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Compare the average daily doses (unit: pills) of the NSAID from Week9 (W9) to W12 between two groups | From W9 to W12 (4 weeks)

SECONDARY OUTCOMES:
Compare the average daily doses (unit: pills) of the NSAID from W5 to W8, and W5 to W12 between two groups | From W5 to W8 (4 weeks), and W5 to W12 (8 weeks)
Compare the changes in the average daily doses (unit: pills) of the NSAID at the 8th and 12th week from baseline between two groups. | At the 8th week from baseline (1 week), and at the 12th week from baseline (1 week)
Compare the percentage changes in the average daily doses (unit: pills) of the NSAID at the 8th and 12th week from baseline between two groups. | At the 8th week from baseline (1 week), and at the 12th week from baseline (1 week)
Compare the days of NSAID consumption from W5 to W8, W9 to W12, and W5 to W12 between two groups. | From W5 to W8 (4 weeks), W9 to W12 (4 weeks), and W5 to W12 (8 weeks)
Compare the changes in WOMAC A1 score (walk-associated pain), WOMAC A, B and C score and patient global assessment (PTGA) at the 4th, 8th and 12th week from baseline between two groups. | At the 4th week from baseline (1 week), at the 8th week from baseline (1 week), and at the 12th week from baseline (1 week)
Compare the changes in clinical observer global assessment (COGA), and scores for activities of daily living (ADL) at the 4th, 8th and 12th week from baseline between two groups. | At the 4th week from baseline (1 week), at the 8th week from baseline (1 week), and at the 12th week from baseline (1 week)

OTHER OUTCOMES:
Incidence of all adverse events (AEs) and serious adverse events (SAEs) | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kun Zheng WANG, Doctor, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality